CLINICAL TRIAL: NCT01466166
Title: Observational Study of the Use of KRYSTEXXA® (Pegloticase) in Adult Hyperuricemic Patients With Gout Refractory to Conventional Therapy
Brief Title: Observational Study of the Use of Pegloticase (KRYSTEXXA®) in Refractory Chronic Gout
Acronym: EyesOnGOUT
Status: Completed | Type: Observational
Sponsor: Horizon Pharma Rheumatology LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: M0401
Record Dates: First submitted 2011-10-28; First posted 2011-11-07 (Estimated); Results first posted 2019-01-11 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2018-06

CONDITIONS: Refractory Chronic Gout
MeSH Terms: interventions — Pegloticase

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pegloticase: Participants received pegloticase 8 mg by intravenous (IV) infusion every 2 weeks for up to 1 year, as prescribed by their treating physician.
  Interventions: Biological: Pegloticase

INTERVENTIONS:
Biological: Pegloticase — Pegloticase 8 mg intravenous every 2 weeks
  Other Names: KRYSTEXXA®

SUMMARY:
The primary purpose of this study is to observe patients being treated with pegloticase in a standard healthcare setting in order to evaluate the frequency and severity of infusion reactions, anaphylaxis and immune complex related events. Additionally, serious adverse events associated with pegloticase therapy will be identified.

DETAILED DESCRIPTION:
This was a Phase 4, multicenter, open-label, single-arm observational study of pegloticase 8 mg administered intravenously every 2 weeks in adult hyperuricemic patients with gout refractory to conventional therapy. Study duration is approximately 63 weeks, including 51 weeks of treatment and 12 weeks of follow-up.

The design of this study follows the FDA-approved Full Prescribing Information for the use of pegloticase and allows for capturing additional data related to the safety and efficacy of pegloticase within the standard healthcare setting.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 18 years or more) with chronic gout refractory to conventional therapy, defined as patients who have failed to normalize SUA and whose signs and symptoms are inadequately controlled with xanthine oxidase inhibitors at the maximum medically appropriate dose, or for whom these drugs are contraindicated.
* Patients who have made the decision, along with their treating physician, to begin treatment with KRYSTEXXA.
* Patients who are willing and able to give informed consent and adhere to visit/protocol schedules.

Exclusion Criteria:

* Glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Non-compensated congestive heart failure
* Pregnancy or breast feeding
* Prior treatment with pegloticase or another recombinant uricase
* Known allergy to urate oxidase
* Prior treatment or concomitant therapy with a polyethylene glycol (PEG)-conjugated drug
* Recipient of an investigational drug within 4 weeks prior to study drug administration or plans to take an investigational agent during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population in this study will be hyperuricemic (serum uric acid (SUA) > 6 mg/dL) adult men and women (age 18 or greater) diagnosed with chronic gout and who are refractory to conventional therapy. Gout refractory to conventional therapy occurs in patients who have failed to normalize SUA and whose signs and symptoms are inadequately controlled with xanthine oxidase inhibitors at the maximum medically appropriate dose or for whom these drugs are contraindicated. To enter this study, the patient and the physician must have decided to begin treatment with KRYSTEXXA.
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2011-11-15 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Nieves, PharmD, Study Director — Horizon Pharma Rheumatology LLC
Locations (67):
- United States (67):
  - Rheumatology Associates, PC, Birmingham, Alabama
  - UAB Rheumatology, Birmingham, Alabama
  - Saadat Ansari, MD, LLC, Huntsville, Alabama
  - Medvin Clinical Research, Covina, California
  - Alliance Clinical Research, LLC, Laguna Hills, California
  - Advanced Medical Research, LLC, Lakewood, California
  - Pacific Arthritis Care Center, Los Angeles, California
  - R Srinivasan, MD, Inc, Monterey Park, California
  - Brigid Freyne, MD, Inc, Murrieta, California
  - Alliance Clinical Research, Poway, California
  - Denver Nephrologists, PC, Denver, Colorado
  - New England Research Associates, LLC, Trumbull, Connecticut
  - Howard University Hospital, Washington D.C., District of Columbia
  - Washington DC Veteran's Affairs Medical Center, Washington D.C., District of Columbia
  - Bay Area Arthritis and Osteoporosis, Brandon, Florida
  - Countryside Arthritis Center, Clearwater, Florida
  - Science and Research Institute, Inc, Jupiter, Florida
  - A & O Research Center, Miami, Florida
  - Arthritis Research of Florida, Inc., Palm Harbor, Florida
  - Family Clinical Trials, LLC, Pembroke Pines, Florida
  - Jedidiah Clinical Research, Tampa, Florida
  - Midtown Medical Center, Tampa, Florida
  - Global Research Partners & Consultants, Inc., Calhoun, Georgia
  - Arthritis Research & Treatment Center, Stockbridge, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Diagnostic Rheumatology and Research PC, Indianapolis, Indiana
  - Physicians' Clinic of Iowa, P.C., Cedar Rapids, Iowa
  - Central Kentucky Research Associates of Kentucky, Mount Sterling, Kentucky
  - Research Integrity, LLC, Owensboro, Kentucky
  - Horizon Research Group of Opelousas, LLC, Eunice, Louisiana
  - Arthritis and Diabetes Clinic, Inc., Monroe, Louisiana
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Klein & Associates MD, PA., Hagerstown, Maryland
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Clinical Pharmacology Study Groups, Worcester, Massachusetts
  - Reliant Medical Group, Inc., Worcester, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Caro Health Plaza, Caro, Michigan
  - Infusion Associates, Grand Rapids, Michigan
  - Justus J. Fiechtner, MD, PC, Lansing, Michigan
  - Shores Rheumatology, PC, Saint Clair Shores, Michigan
  - Saint Paul Rheumatology, PA, Eagan, Minnesota
  - Kansas City Internal Medicine, Kansas City, Missouri
  - Arthritis Medical Clinic, Las Vegas, Nevada
  - Rheumatology Associates of North Jersey, Teaneck, New Jersey
  - Rheumatology Associates of Long Island, Smithtown, New York
  - NorthEast Rheumatology, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Physicians East, PA, Greenville, North Carolina
  - Shanahan Rheumatology and Immunotherapy, PLLC, Raleigh, North Carolina
  - Specialty Medical Clinic and Research Center, Sanford, North Carolina
  - Southern Ohio Rheumatology, Portsmouth, Ohio
  - Keystone Pain Institute, Ilumina Clinical Associates, Altoona, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Low Country Rheumatology, Charleston, South Carolina
  - Acme Research L.L.C., Orangeburg, South Carolina
  - Ramesh C. Gupta, M.D., Memphis, Tennessee
  - Austin Regional Clinic, Austin, Texas
  - Dr. Raj Marwah, El Paso, Texas
  - Diagnostic Clinic of Houston, Houston, Texas
  - Rheumatic Disease Clinical Research Center, Houston, Texas
  - Arthritis Clinic of Northern Virginia, P.C., Arlington, Virginia
  - Arthritis & Osteoporosis Center of North Virginia, Manassas, Virginia
  - Sentara Rheumatology Specialists, Norfolk, Virginia
  - Apex Clinical Research, Kennewick, Washington
  - Mountain State Clinical Research, Clarksburg, West Virginia
  - Rheumatic Disease Center, LLP, Glendale, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sundy JS, Baraf HS, Yood RA, Edwards NL, Gutierrez-Urena SR, Treadwell EL, Vazquez-Mellado J, White WB, Lipsky PE, Horowitz Z, Huang W, Maroli AN, Waltrip RW 2nd, Hamburger SA, Becker MA. Efficacy and tolerability of pegloticase for the treatment of chronic gout in patients refractory to conventional treatment: two randomized controlled trials. JAMA. 2011 Aug 17;306(7):711-20. doi: 10.1001/jama.2011.1169. PMID 21846852
- See also: Related Info — https://www.krystexxa.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 249 patients were screened at 66 of 112 activated clinical sites in the United States; 61 (24.5%) of the 249 patients were screen failures and 188 were enrolled.
Period: Overall Study
Arm/Group | Pegloticase
Started | 188
Received Treatment | 188
Completed 24 Weeks of Treatment | 55
Completed (Patients completed the treatment phase of the study (on study for 52 weeks)) | 25
Not Completed | 163
Not completed — Death | 1
Not completed — Lost to Follow-up | 7
Not completed — Infusion Reaction (IR) | 27
Not completed — Adverse Event (Other than IR) | 11
Not completed — Elevated Serum Uric Acid | 78
Not completed — Withdrawal by Subject | 13
Not completed — Sponsor Decision | 4
Not completed — Protocol Violation/Noncompliance | 2
Not completed — Other | 20

BASELINE CHARACTERISTICS:
Arm/Group | Pegloticase
Number analyzed (Participants) | 188
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.32 (13.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 169
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 168
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 131
  Asian | 16
  Black or African American | 30
  Native Hawaiian or Pacific Islander | 1
  American Indian or Alaskan Native | 2
  Other | 8
Baseline Serum Uric Acid [Mean (Standard Deviation); unit: mg/dL] — Population: Participants with available data
  mg/dL
    number analyzed (Participants) | 185
    (all) | 9.03 (2.29)
Duration Since Initial Gout Diagnosis [Mean (Standard Deviation); unit: years] | 15.54 (10.36)
Number of Gout Flares in Last 6 Months [Mean (Standard Deviation); unit: flares] | 7.60 (12.17)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Infusion Reactions
Description: Infusion reactions were defined as adverse events (AEs) or clusters of events, not attributable to another cause that occurred during or within 2 hours after the infusion of pegloticase. Any other case that occurred outside of the 2-hour window was categorized per Investigator discretion.
Time Frame: 52 weeks
Population: The intent-to-treat population included all enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Pegloticase
Number analyzed (Participants) | 188
Participants | 42

2. Primary Outcome: Number of Participants With Anaphylaxis
Description: Anaphylaxis was defined using the National Institute of Allergy and Infectious Disease/Food Allergy and Anaphylaxis Network (NIAID/FAAN) criteria: Acute onset of an illness (minutes to several hours) with involvement of the skin, mucosal tissue, or both (e.g., generalized hives; pruritus or flushing; swollen lips, tongue, or uvula), and at least 1 of the following:
  1. Respiratory compromise (e.g., dyspnea, wheeze-bronchospasm, stridor, reduced peak expiratory flow, hypoxemia).
  2. Reduced blood pressure (i.e., systolic blood pressure < 90 mm Hg or greater than 30% decrease from that patient's baseline) or associated symptoms of end-organ failure (e.g., hypotonia [collapse], syncope, incontinence).
Time Frame: 52 weeks
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Pegloticase
Number analyzed (Participants) | 188
Participants | 5

3. Primary Outcome: Number of Participants With Immune Complex-related Events
Description: Immune complex-related events were defined as any presumptive immune complex-related disorders that were confirmed by an appropriate investigation of the event and of complement markers (C3 and C4 levels). Clinical manifestations could have included skin rash, arthralgia, arthritis, proteinuria, serum sickness, and cryoglobulinemia.
Time Frame: From first dose of study drug to the end of the 12-week follow-up period (63 weeks).
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Pegloticase
Number analyzed (Participants) | 188
Participants | 3

4. Secondary Outcome: Percentage of Participants With Normalization of Serum Uric Acid at Week 24 and Week 52
Description: Normalization of serum uric acid was defined as serum uric acid value less than 6 mg/dL.
Time Frame: Week 24 and week 52
Population: Participants with missing values at week 24 or 52 are counted as not achieving normalization
Measure: Number; unit: percentage of participants
Arm/Group | Pegloticase
Number analyzed (Participants) | 188
percentage of participants
  Week 24 | 27.7
  Week 52 | 12.2

5. Secondary Outcome: Change From Baseline in Number of Gout Flares
Description: The number of gout flares occurring in the 2 weeks prior to each visit. Baseline number of flares was calculated as the average number of flares that occurred in the 6-month baseline period divided by 12 weeks.
Time Frame: Baseline, week 24 and week 48
Population: Enrolled participants with a value at baseline and each time point
Measure: Mean (Standard Deviation); unit: flares
Arm/Group | Pegloticase
Number analyzed (Participants) | 188
flares
  Week 24: number analyzed (Participants) | 46
  Week 24 | -0.83 (0.88)
  Week 48: number analyzed (Participants) | 26
  Week 48 | -1.00 (0.89)

6. Secondary Outcome: Number of Swollen Joints Over Time
Time Frame: Baseline and weeks 24 and 52
Population: Enrolled participants with available data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Pegloticase
Number analyzed (Participants) | 188
swollen joints
  Baseline: number analyzed (Participants) | 186
  Baseline | 8.60 (10.847)
  Week 24: number analyzed (Participants) | 42
  Week 24 | 4.05 (7.241)
  Week 52: number analyzed (Participants) | 24
  Week 52 | 1.46 (3.336)

7. Secondary Outcome: Number of Tender Joints Over Time
Time Frame: Baseline and weeks 24 and 52
Population: Enrolled participants with available data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Pegloticase
Number analyzed (Participants) | 188
tender joints
  Baseline: number analyzed (Participants) | 186
  Baseline | 9.33 (11.715)
  Week 24: number analyzed (Participants) | 42
  Week 24 | 2.38 (5.539)
  Week 52: number analyzed (Participants) | 24
  Week 52 | 0.79 (1.318)

8. Secondary Outcome: Number of Palpable Tophi Over Time
Description: Gout tophi are nodular deposits of urate crystals and inflammatory cells in joints, soft tissues, bones, and in some organs.
Time Frame: Baseline and weeks 24 and 52
Population: Enrolled participants with available data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: tophi
Arm/Group | Pegloticase
Number analyzed (Participants) | 188
tophi
  Baseline: number analyzed (Participants) | 161
  Baseline | 13.58 (18.999)
  Week 24: number analyzed (Participants) | 33
  Week 24 | 5.70 (5.643)
  Week 52: number analyzed (Participants) | 19
  Week 52 | 3.68 (3.038)

ADVERSE EVENTS:
Time Frame: From first dose of study drug to the end of the 12-week follow-up period (63 weeks).
Arm/Group | Pegloticase
All-Cause Mortality (participants affected / at risk) | 3/188
Serious Adverse Events (participants affected / at risk) | 31/188
Other Adverse Events (participants affected / at risk) | 130/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pegloticase (N=188)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 2
Coronary artery disease (Cardiac disorders) | 1
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Anaphylaxis (Immune system disorders) | 5
Drug hypersensitivity (Immune system disorders) | 3
Cellulitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Gout (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 2
Renal failure (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 4
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pegloticase (N=188)
Drug hypersensitivity (Immune system disorders) | 11
Gout (Metabolism and nutrition disorders) | 126

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Horizon requests that any investigator/institution that plans on presenting/publishing results provide written notification of their request 60 days prior to their presentation/publication. Horizon requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Horizon needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2011-07-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT01466166/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-25): https://cdn.clinicaltrials.gov/large-docs/66/NCT01466166/SAP_001.pdf